CLINICAL TRIAL: NCT02204800
Title: Active Surveillance of the Small Renal Mass: An Integrated Biomarker Trial
Brief Title: Active Surveillance of the Small Renal Mass
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1312013110; Yale Department of Urology (Other: Yale Department of Urology)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Small Renal Mass, Kidney Cancer
Keywords: Tumor growth rate in maximal dimension, biomarker assessment based on driver gene alterations (specifically CRG)
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Small clear cell renal tumors (Wild Type): No specific chromatin remodeling gene (CRG) alteration
- Small clear cell renal tumors (Mutant): Specific chromatin remodeling gene (CRG) alteration

SUMMARY:
Active surveillance in kidney cancer involves closely observing the tumor with periodic imaging studies rather than immediately proceeding to an invasive treatment. This does not mean that the tumor is ignored or that future treatment is not necessary, rather it means the tumor does not require treatment at this time. On active surveillance, a tumor is closely monitored without treatment, however if the tumor changes and reaches a predefined threshold that your physician no longer considers safe, your physician will strongly encourage treatment.

DETAILED DESCRIPTION:
While some patients with small kidney tumors may require eventual treatment, most do not. Therefore, the American Urologic Association considers active surveillance an acceptable treatment strategy. This protocol is a prospective study of active surveillance for small clear cell kidney tumors (the most common type of kidney tumor) and is designed to identify if there are predictive markers that may help identify which patients are unlikely to require surgical treatment. Predictive markers are measurable characteristics that may predict the future behavior of a tumor. There are currently no available predictive markers that can help identify which tumors are not destined to require treatment. Such a marker may be useful to increase the use of active surveillance by informing patients with small renal tumors that immediate treatment may be considered overtreatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Life expectancy >3 years (by physician estimate)
* Measurable, solid renal neoplasm, 1.0 -2.7 cm in size and visible on ultrasound
* Clear cell renal cell carcinoma histology
* Renal tumor diagnosed within 6 months
* Recent biopsy (<6 weeks) performed, if performed at an outside institution, there must be sufficient material for biomarker analysis
* No evidence of vascular invasion or regional nodal/distant disease
* Renal tumor that is able to be managed with upfront surgery
* Adequate organ function (Hemoglobin > 9, Absolute neutrophil count (ANC) ≥ 1500/μL Platelets ≥ 100,000/μL, AST and ALT ≤3.0 upper limit of normal (ULN), total bilirubin ≤ ULN, eGFR ≥ 30
* Good Performance status (ECOG ≤2)
* Understanding and willingness to provide consent

Exclusion Criteria:

* History of a hereditary renal cancer syndrome
* Tumor >2.7 cm, stages T1b-T4
* Life expectancy <3 years
* Presence of an active, untreated, metastatic non-renal malignancy
* Uncontrolled medical illness including infections, hypertension, arrhythmias, heart failure, or myocardial infarction within 6 months that would predispose to immediate surgical therapy
* Medical contraindication to upfront surgical management of renal mass
* History of bleeding diathesis or recent bleeding episode that would prevent surgical resection
* Unwillingness to undergo monitoring and imaging studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a trial of active surveillance in patients with a solitary, small (1.0-2.7 cm) renal mass.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Tumor growth rate | 36 months
  Tumor growth rate is being measured in centimeters/year

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shuch, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Smilow Cancer Center, New Haven, Connecticut, United States